CLINICAL TRIAL: NCT06599294
Title: Accuracy of Intraoral Photogrammetry Scanner (IPS) in Complete Arch Digital Implant Impression: an in Vivo Prospective Comparative Study
Brief Title: Accuracy of Intraoral Photogrammetry Scanner in Complete Arch Digital Implant Impression
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Collaborators: Assiut University (Other)
Responsible Party: Principal Investigator, Doaa Adel Salah Khattab, Associate Professor, Ain Shams University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 112899
Record Dates: First submitted 2024-09-07; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-07

CONDITIONS: Dental Implant
Keywords: Digital; photogrammetry; Intra oral scanner

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intraoral photogrammetry scanning (Experimental)
  Interventions: Procedure: Digital scanning; Procedure: Two digital impressions will be recorded, one with a conventional intra-oral scanner and another one with an intra-oral photogrammetry scanner.
- Intra oral scanning (Active Comparator)
  Interventions: Procedure: Digital scanning; Procedure: Two digital impressions will be recorded, one with a conventional intra-oral scanner and another one with an intra-oral photogrammetry scanner.

INTERVENTIONS:
Procedure: Digital scanning — . For each patient three digital files will be obtained: One reference scan, one conventional IOS scan, and one IPS scan. All the STL files will be imported to dental CAD software, and scan bodies will be converted to implant multi-unit ti-base using a digital library. The updated STL files will be imported to inspection software Mimics for trueness assessments. The three-dimensional discrepancy between 2 STL files will be evaluated in terms of linear and angular deviation. A central point & central axis of the virtual MUA ti-base was used for deviation measurements. Linear deviations will be assessed for each MUA tibase on the three-space axis (X longitudinal, Y lateral, and Z vertical) using the center of the ti-base heads for the deviation measurement. Angular deviations were assessed as the angles formed by the two lines passing perpendicularly through the centers of the test image and the reference image of each ti-base.
Procedure: Two digital impressions will be recorded, one with a conventional intra-oral scanner and another one with an intra-oral photogrammetry scanner. — . For each patient three digital files will be obtained: One reference scan, one conventional IOS scan, and one IPS scan. All the STL files will be imported to dental CAD software, and scan bodies will be converted to implant multi-unit ti-base using a digital library. The updated STL files will be imported to inspection software Mimics for trueness assessments. The three-dimensional discrepancy between 2 STL files will be evaluated in terms of linear and angular deviation. A central point & central axis of the virtual MUA ti-base was used for deviation measurements. Linear deviations will be assessed for each MUA tibase on the three-space axis (X longitudinal, Y lateral, and Z vertical) using the center of the ti-base heads for the deviation measurement. Angular deviations were assessed as the angles formed by the two lines passing perpendicularly through the centers of the test image and the reference image of each ti-base.

SUMMARY:
Intra oral scanning can perform a full digital workflow right on the patient's mouth. Recently an intra-oral photogrammetry scanner has been introduced in the market that can make intra-oral tissue scanning in addition to a built-in photogrammetry technology so that it can capture fixture locations through special intra-oral scan flags.

DETAILED DESCRIPTION:
Intraoral scanning had several advantages to intraoral direct scanning, including less storage and transportation needs, faster scanning times, and increased patient comfort. The intraoral scan bodies are used as digital fixture locators when using IOSs for implant impressions.

Photogrammetry is the science and technology of obtaining reliable information about physical objects through the process of recording, measuring, and interpreting photographic images and patterns of electromagnetic radiant imagery. The utilization of photogrammetry in the dental field leads to exclusion of intraoral dental and gingival anatomies while scanning the implant coordinates. In addition, no need for stitching during full arch implant scanning which is reflected in the trueness and precision of the scanned object. Exclusion of unstable mucosa during scanning and avoidance of stitching make the passive seating of implant prosthesis a more predictable procedure especially when compared with intra-oral scanning only.

Up to this moment, all photogrammetry systems available in the market are considered extraoral systems that require an additional impression for soft tissue capture whether conventional or digital. Recently an intra-oral photogrammetry scanner (IPS) has been introduced in the market that can make intra-oral tissue scanning in addition to a built-in photogrammetry technology so that it can capture fixture locations through special intra-oral scan flags.

ELIGIBILITY:
Inclusion Criteria:

* participants had received 4-6 implants in 1 edentulous arch.
* Participants had received 1-piece implant-supported complete-arch fixed dental prostheses.

Exclusion Criteria:

* Systemic conditions as diabetes.
* Osteoporosis patients.
* Immunocompromised patients.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-06-20 (Actual); Primary Completion 2024-08-10 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
Degree of Trueness | 4 months following implant insertion
  The clinical performance of conventional intraoral scanners (IOS) and intraoral photogrammetry scanners (IPS) for each patient enrolled in the study with a paired comparison of the deviation differences

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry Ain Shams University, Cairo, Abbassia, Egypt

IPD SHARING:
Plan to Share IPD: No